CLINICAL TRIAL: NCT01271465
Title: mRNA and microRNA Profiles in Renal Transplant at the Time of Organ Reperfusion
Brief Title: Analysis of Donor Biopsy Tissue Samples at the Time of Kidney Transplant
Status: Completed | Type: Observational
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: Qatar National Research Fund (Other)
Responsible Party: Sponsor
Other Study IDs: 1004010988
Record Dates: First submitted 2011-01-05; First posted 2011-01-06 (Estimated); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Kidney Transplantation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, urine, and kidney tissue will be analyzed for mRNA and microRNA expression of pro-inflammatory genes.

INTERVENTIONS:
Procedure: Kidney Biopsy — biopsy of transplant kidney

SUMMARY:
The purpose of this study is to see if substances measured in a small piece of the donor organ predicts how well the organ will function in the recipient after transplant. We will be testing blood, urine, and biopsy tissue samples in this study. The research team will be looking at different risk factors in the donor organ that predict how well the kidney will do in the recipient.

DETAILED DESCRIPTION:
Background:

Early post-transplant kidney function can be attributed to inherent donor characteristics, damage from storage, and perioperative events and recipients factors. The incidence of severe injury to the transplant kidneys is 10-25% in the early post-transplant period. In addition, milder forms of early transplant kidney injury can impact on long term allograft function. Severe transplant kidney injury in the immediate post-transplant period has been hypothesized to be associated with higher rates of rejection.

Hypothesis:

In the current investigation, we would like to test the hypotheses that 1) mRNA and microRNA expression of proinflammatory genes in donor tissues is a risk factor for development of early kidney transplant dysfunction and 2) early inflammatory mRNA and microRNA expression in the allograft is associated with subsequent activation of cell mediated immunity as evidenced by increased incidence of acute rejection episodes and increased expression of cell mediated immunity genes during the first year post-transplant.

Aims:

Aim 1: Test the association between proinflammatory mRNA and microRNA expression in donor samples and subsequent development of early organ dysfunction in the immediate period following transplantation.

Aim 2: Test the association of mRNA and microRNA expression of proinflammatory mediators in the transplanted organ in the immediate pre and post-reperfusion period with subsequent incidence of acute rejection and expression of genes involved in cell mediated immunity.

ELIGIBILITY:
Inclusion Criteria:

* Males and females <80 years of age for kidney
* Recipients of single abdominal organ transplant
* Ability to provide written informed consent
* Donor blood and kidney biopsy tissues specimens are collected at the time of transplantation

Exclusion Criteria:

* Need for combined organ transplantation.
* Inability or unwillingness of a participant or legal guardian to provide written informed consent
* Clinical evidence of systemic bacterial infection in the recipient at the time of transplantation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Renal allograft recipients are generally in good health and many return to work by three months post-transplant.
  However, they are maintained on immunosuppressive medications to maintain the function of the transplanted kidney.
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2010-09 (Actual); Primary Completion 2021-09-18 (Actual); Study Completion 2021-09-18 (Actual)

PRIMARY OUTCOMES:
Incidence of early organ dysfunction, defined by standard criteria for each organ defined as the need for dialysis within 7 days after transplant and incidence of biopsy proven acute cellular rejection within 12 months of transplant | 7 days and 12 months, respectively

SECONDARY OUTCOMES:
Serum Creatinine | 24 months
  Correlation between proinflammatory mediators at the time of transplantation and renal function as measured by serum creatinine
Incidence of chronic allograft nephropathy | 24 months
  Correlation between proinflammatory mediators at the time of transplantation and incidence of chronic allograft nephropathy

CONTACTS AND LOCATIONS:
Overall Officials: Samuel Sultan, MD, Principal Investigator — Weill Cornell Medicine/Department of Surgery
Locations (1):
- Weill Cornell Medical College, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided